CLINICAL TRIAL: NCT03709576
Title: A Phase II Study of Pevonedistat (MLN4924, TAK924) and Azacitidine as Maintenance Therapy After Allogeneic Stem Cell Transplantation for Non-Remission Acute Myelogenous Leukemia
Brief Title: Pevonedistat and Azacitidine as Maintenance Therapy After Allogeneic Stem Cell Transplantation for Non-Remission AML
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding pulled
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Takeda (Industry)
Responsible Party: Principal Investigator, Shin Mineishi, Professor and Director, Blood and Marrow Transplant Program, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSCI 17-056
Record Dates: First submitted 2018-07-26; First posted 2018-10-17 (Actual); Results first posted 2020-10-29 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pevonedistat; Transplantation; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pevonedistat and Azacitidine (Experimental): The study period is from the start of study treatment, cycle 1 day 1 until 28 days after the last treatment dose. (Cycle 5 day 9). Treatment will be continued until cycle 5 is completed or the study is terminated for the patient. The cycles will be repeated every 28 days. Cycle 1 Day 1 of study treatment will be between day +30 and day +45 post-transplant. Each 28-day cycle is comprised of Pevonedistat at 20 mg/m2 IV infusion over 1 hour on days 1, 3 and 5 and Azacitidine at 25 mg/m2 IV infusion over 30 minutes on days 1, 2, 3, 4, 5, 8 and 9. The drugs can be administered either through a central catheter or a peripheral line.
  Interventions: Drug: Pevonedistat; Procedure: transplant; Drug: Azacitidine

INTERVENTIONS:
Drug: Pevonedistat — To assess the toxicity and efficacy of a combination of Pevonedistat and Azacitidine as post allogeneic hematopoietic stem cell transplant maintenance therapy for non-remission AML.
Procedure: transplant — Although hematopoietic stem cell transplantation (HSCT) is curative for many patients with AML, AML in relapse at the time of transplant is still a major challenge with low rates of leukemia-free survival even with an intensive myeloablative conditioning.
Drug: Azacitidine — To assess the toxicity and efficacy of a combination of Pevonedistat and Azacitidine as post allogeneic hematopoietic stem cell transplant maintenance therapy for non-remission AML.

SUMMARY:
This research is being done to find out the toxicity and efficacy of a combination of Pevonedistat and Azacitidine as post allogeneic hematopoietic stem cell transplant maintenance therapy for non-remission AML and to see the overall diseases free survival, relapse, and GVHD after treatment.

DETAILED DESCRIPTION:
In preclinical studies Pevonedistat has shown significant single agent activity against mouse xenograft models of AML cell Line HL-60. Also this effect seemed to be synergistically enhanced by combining it with Azacitidine. In clinical arena, Pevonedistat has shown single agent activity in heavily pretreated patients with AML. In Study C15003, responses (complete responses [CRs] and partial responses [PRs]) were observed in a variety of patient settings, including post allogeneic transplant, therapy-related AML, and primary refractory AML, although some of the responses were of relatively short duration. Study C15009 is an ongoing phase 1b study evaluating the MTD of Pevonedistat on Days 1, 3, and 5 in combination with 75 mg/m2 Azacitidine (administered on a 5-on/2-off [weekend]/2-on schedule) in a 28-day treatment cycle in patients 60 years of age or older with treatment naïve AML who are unlikely to benefit from standard induction therapy. As of 22 June 2017, enrollment had completed and 15 patients remained on study. As of 22 January 2017, preliminary data are available for 64 patients enrolled in the study who received at least 1 dose of Pevonedistat in combination with Azacitidine; these patients had completed a total of approximately 360 cycles, with a median of 4 cycles of treatment In the dose escalation cohorts, 6 patients received 20 mg/m2 Pevonedistat, and 3 patients received 30 mg/m2. The most common events (reported by ≥ 25% of patients) were constipation (45%), nausea (42%), fatigue (39%), anemia (34%), febrile neutropenia (30%), decreased appetite (28%), and thrombocytopenia (27%). The MTD in this study was determined to be 20 mg/m2 Pevonedistat given on Days 1, 3, and 5, in combination with 75 mg/m2 Azacitidine given on Days 1 through 5, 8, and 9, in 28 day treatment cycles. A total of 45 (70%) patients experienced at least 1 SAE A total of 14 SAEs were reported for more than 1 patient, including: febrile neutropenia (16 patients); pneumonia (8 patients); pyrexia (4 patients); AML and sepsis (3 patients); and acute myocardial infarction, cellulitis, diverticulitis, dyspnea, embolism, hypoxia, mental status changes, multi-organ failure, and transaminase increased (2 patients each). A total of 19 patients treated with Pevonedistat (either 20 mg/m2 or 30 mg/m2), discontinued from Study participation because of a TEAE. No other events leading to discontinuation were assessed by study investigators as at least possibly related to study drug treatment. 11 on-study deaths had been reported; none assessed as related to study treatment. A total of 31 patients experienced PR or better. Eighteen patients had a best response of CR, 4 patients had a best response of CRi, and 9 patients had a best response of PR. One patient in the 30 mg/m2 dose level group achieved a CR; all other responses occurred in patients treated with 20 mg/m2.

The following studies are currently enrolling.

* Study 2001: A Phase 2, randomized, controlled Open-Label Clinical study of the efficacy and safety of Pevonedistat plus Azacitidine versus single-agent Azacitidine in patients with higher-risk myelodysplastic syndromes, chronic myelomonocytic leukemia and low-blast acute myelogenous leukemia.
* Study 1012: A phase 1/1b, Open-label Study of Pevonedistat (MLN4924, TAK-924) as Single Agent and in Combination with Azacitidine in adult East Asian patients with acute myeloid leukemia or myelodysplastic syndromes

Hence owing to the current knowledge of clinical and preclinical experience with Azacitidine and Pevonedistat alone and in combination, this combination appears feasible for testing in patients post-transplant with at very high risk of relapse.

The Investigator proposes a study using a combination of Pevonedistat and Azacitidine for maintenance therapy after allogeneic HSCT for non-remission. Patients will receive up to five 28 day cycles of the investigational maintenance therapy. Maintenance therapy will begin between days +30 to +45 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years (or age of majority at participating site, whichever is greater) and ≤ 70 years.
2. Non-remission AML at the time of transplant proven via bone marrow aspiration and/or biopsy.

   o"Not in remission" is defined as "greater than 5.0% bone marrow blasts by aspirate morphology," as determined by a bone marrow aspirate obtained within 2 weeks of study registration.
   * For primary induction failure patients: Patients must have failed at least 2 induction regimens.
   * For patients with relapsed disease: Patients who relapse more than 6 months after preceding remission must fail at least one reinduction regimen to be eligible. For patients in whom the preceding remission is equal to or shorter than 6 months duration, no re-induction regimen is required to qualify for this protocol.
   * If the pre-transplant bone marrow aspirate and biopsy are hypo plastic (less than 10% cellularity), and blast percentages cannot be determined, the patient is eligible if the preceding bone marrow met the above criteria.
   * Patients with peripheral circulating blasts or patients with extramedullary leukemia are eligible if bone marrow aspirate and biopsy meets the above criteria.
3. Karnofsky Performance Scale (KPS) above or equal to 70%
4. Clinical laboratory values within the following parameters (repeat if more than 3 days before the first dose):

   1. Creatinine clearance ≥ 50 mL/min
   2. Hemoglobin > 8 g/dL. Patients may be transfused to achieve this value.
   3. White blood cell (WBC) count < 50,000/µL before administration of Pevonedistat on Cycle 1 Day 1. Note: Hydroxyurea may be used to control the level of circulating leukemic blast cell counts to not lower than 10,000/µL during the study.
   4. LFTs (ALT, AST) equal or less than 2.5 times upper limit of normal value.
   5. Bilirubin ≤ x 1.5 ULN limit
5. Female patients who:

   * Are postmenopausal (see Appendix for definition) for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR

   If they are of childbearing potential:
   * Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception (see Appendix), at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

   Male patients, even if surgically sterilized (i.e., status post vasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (female and male condoms should not be used together), or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
6. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Treatment with any investigational products within 21 days of study registration.
2. Known hypersensitivity to Azacitidine.
3. Active uncontrolled infections or severe infectious disease, such as severe pneumonia, meningitis, or septicemia.
4. Known central nervous system (CNS) involvement.
5. Known human immunodeficiency virus (HIV) positivity.
6. Known hepatitis B surface antigen-positive, or known active hepatitis C infection.

   * Note: Patients who have isolated positive hepatitis B core antibody (ie, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
7. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures
8. Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during study period.
9. Diagnosed or treated for another malignancy within 2 years before randomization or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non- melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection.
10. Life-threatening illness unrelated to cancer.
11. Patients with uncontrolled coagulopathy or bleeding disorder.
12. Known hepatic cirrhosis or severe pre-existing hepatic impairment
13. Known cardiopulmonary disease defined as:

    * Unstable angina;
    * Congestive heart failure (New York Heart Association [NYHA] Class III or IV; see appendix);
    * Myocardial infarction (MI) within 6 months prior to first dose (patients who had ischemic heart disease such as a (ACS), MI, and/or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll);
    * Cardiomyopathy;
    * Clinically significant arrhythmia:

      1. History of polymorphic ventricular fibrillation or torsade de pointes,
      2. Permanent atrial fibrillation [a fib], defined as continuous a fib for ≥ 6 months,
      3. Persistent a fib, defined as sustained a fib lasting > 7 days and/or requiring cardioversion in the 4 weeks before screening,
      4. Grade 3 a fib defined as symptomatic and incompletely controlled medically, or controlled with device (e.g. pacemaker), or ablation and
      5. Patients with paroxysmal a fib or < Gr 3 a fib for period of at least 6 months are permitted to enroll provided that their rate is controlled on a stable regimen.
    * Implantable cardioverter defibrillator;
    * Moderate to severe aortic and/or mitral stenosis or other valvulopathy (ongoing);
    * Pulmonary hypertension
14. Uncontrolled high blood pressure (i.e., systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg).
15. Prolonged rate corrected QT (QTc) interval ≥ 500 msec, calculated according to institutional guidelines.
16. Left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram or radionuclide angiography.
17. Known moderate to severe chronic obstructive pulmonary disease, interstitial lung disease, and pulmonary fibrosis.
18. Systemic antineoplastic therapy or radiotherapy for other malignant conditions within 14 days before the first dose of any study drug, except for hydroxyurea.
19. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.
20. Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).
21. Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s).
22. Patients who need to use clinically significant CYP3A enzyme inducers (listed on Appendix A)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shin Mineishi, MD, Principal Investigator — Penn State Cancer Institute (Hershey Medical Center)
Locations (1):
- Penn State Hershey Medical Center: Penn State Cancer Institute, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Sierra J, Storer B, Hansen JA, Bjerke JW, Martin PJ, Petersdorf EW, Appelbaum FR, Bryant E, Chauncey TR, Sale G, Sanders JE, Storb R, Sullivan KM, Anasetti C. Transplantation of marrow cells from unrelated donors for treatment of high-risk acute leukemia: the effect of leukemic burden, donor HLA-matching, and marrow cell dose. Blood. 1997 Jun 1;89(11):4226-35. PMID 9166868
- [Background] Giralt S, Estey E, Albitar M, van Besien K, Rondon G, Anderlini P, O'Brien S, Khouri I, Gajewski J, Mehra R, Claxton D, Andersson B, Beran M, Przepiorka D, Koller C, Kornblau S, Korbling M, Keating M, Kantarjian H, Champlin R. Engraftment of allogeneic hematopoietic progenitor cells with purine analog-containing chemotherapy: harnessing graft-versus-leukemia without myeloablative therapy. Blood. 1997 Jun 15;89(12):4531-6. PMID 9192777
- [Background] Saito T, Kanda Y, Kami M, Kato K, Shoji N, Kanai S, Ohnishi T, Kawano Y, Nakai K, Ogasawara T, Matsubara H, Makimoto A, Tanosaki R, Tobinai K, Wakasugi H, Takaue Y, Mineishi S. Therapeutic potential of a reduced-intensity preparative regimen for allogeneic transplantation with cladribine, busulfan, and antithymocyte globulin against advanced/refractory acute leukemia/lymphoma. Clin Cancer Res. 2002 Apr;8(4):1014-20. PMID 11948108
- [Background] Kassim AA, Chinratanalab W, Ferrara JL, Mineishi S. Reduced-intensity allogeneic hematopoietic stem cell transplantation for acute leukemias: 'what is the best recipe?'. Bone Marrow Transplant. 2005 Oct;36(7):565-74. doi: 10.1038/sj.bmt.1705075. PMID 15995714
- [Background] Slavin S, Nagler A, Naparstek E, Kapelushnik Y, Aker M, Cividalli G, Varadi G, Kirschbaum M, Ackerstein A, Samuel S, Amar A, Brautbar C, Ben-Tal O, Eldor A, Or R. Nonmyeloablative stem cell transplantation and cell therapy as an alternative to conventional bone marrow transplantation with lethal cytoreduction for the treatment of malignant and nonmalignant hematologic diseases. Blood. 1998 Feb 1;91(3):756-63. PMID 9446633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Penn State Milton S. Hershey Medical Center from 18 July 2018 through 17 October 2019
Pre-assignment Details: One subject was excluded due to progression of disease prior to enrollment
Groups:
- Pevonedistat and Azacitidine: The study period is from the start of study treatment, cycle 1 day 1 until 28 days after the last treatment dose. (Cycle 5 day 9). Treatment will be continued until cycle 5 is completed or the study is terminated for the patient. The cycles will be repeated every 28 days. Cycle 1 Day 1 of study treatment will be between day +30 and day +45 post-transplant. Each 28-day cycle is comprised of Pevonedistat at 20 mg/m2 IV infusion over 1 hour on days 1, 3 and 5 and Azacitidine at 25 mg/m2 IV infusion over 30 minutes on days 1, 2, 3, 4, 5, 8 and 9. The drugs can be administered either through a central catheter or a peripheral line.
  Pevonedistat: To assess the toxicity and efficacy of a combination of Pevonedistat and Azacitidine as post allogeneic hematopoietic stem cell transplant maintenance therapy for non-remission AML.
  transplant: Although hematopoietic stem cell transplantation (HSCT) is curative for many patients with AML, AML in relapse at the time of transplant is still a
Period: Overall Study
Arm/Group | Pevonedistat and Azacitidine
Started | 3
Completed | 2
Not Completed | 1
Not completed — progression prior to enrollment | 1

BASELINE CHARACTERISTICS:
Population: This research is being done to find out the toxicity and efficacy of a combination of Pevonedistat and Azacitidine as post allogeneic hematopoietic stem cell transplant maintenance therapy for non-remission AML and to see the overall diseases free survival, relapse, and GVHD after treatment
Groups:
- Pevonedistat and Azacitidine: The study period is from the start of study treatment, cycle 1 day 1 until 28 days after the last treatment dose. (Cycle 5 day 9). Treatment will be continued until cycle 5 is completed or the study is terminated for the patient. The cycles will be repeated every 28 days. Cycle 1 Day 1 of study treatment will be between day +30 and day +45 post-transplant. Each 28-day cycle is comprised of Pevonedistat at 20 mg/m2 IV infusion over 1 hour on days 1, 3 and 5 and Azacitidine at 25 mg/m2 IV infusion over 30 minutes on days 1, 2, 3, 4, 5, 8 and 9.
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (4.9)
Sex/Gender, Customized [Count of Participants; unit: Participants] | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: One Year Overall Survival Assessed by the Kaplan-Meier Plots
Description: One year overall survival assess by Kaplan Meier Plots
Time Frame: 1 year
Population: Data could not be reported in the data table as the data were not collected due to study early termination.
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 0

2. Primary Outcome: To Assess the Toxicity and Efficacy of a Combination of Pevonedistat and Azacitidine as Post Allogeneic Hematopoietic Stem Cell Transplant Maintenance Therapy for Non-remission AML.
Description: Toxicity and efficacy unable to be determined as trial was closed by the sponsor prior to meeting this objective.
Time Frame: not analyzed
Population: Data could not be reported in the data table as the data were not collected due to study early termination.
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 0

3. Primary Outcome: Toxicity Related to Pevonedistat
Description: Toxicity related to Pevonedistat unable to be determined as trial was closed by sponsor prior to meeting this objective
Time Frame: not analyzed
Population: Data could not be reported in the data table as the data were not collected due to study early termination.
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 0

4. Secondary Outcome: To Assess the Overall Disease Free Survival, Relapse, and GVHD After the Above Noted Treatment
Description: overall disease free survival, relapse and GVHD unable to be determined as trial was closed by the sponsor prior to meeting this objective
Time Frame: not analyzed
Population: Data could not be reported in the data table as the data were not collected due to study early termination.
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 0

5. Secondary Outcome: One-year Disease-free Survival
Description: One-year disease-free survival unable to be determined as trail was closed by the sponsor prior to meeting this endpoint
Time Frame: not analyzed
Population: Data could not be reported in the data table as the data were not collected due to study early termination.
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 0

6. Secondary Outcome: Cumulative Incidence of Relapse at 2 Years
Description: Cumulative incidence of relapse at 2 years unable to be determined as trial was closed by the sponsor prior to meeting this objective
Time Frame: not analyzed
Population: Data could not be reported in the data table as the data were not collected due to study early termination.
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 0

7. Secondary Outcome: Two-year and Five-year Disease-free and Overall Survival
Description: Two-year and five-year disease-free and overall survival unable to be determined as trial was closed by the sponsor prior to meeting this objective
Time Frame: not analyzed
Population: Data could not be reported in the data table as the data were not collected due to study early termination.
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 0

8. Secondary Outcome: Treatment Related Mortality/Morbidity
Description: Treatment related mortality/morbidity unable to be determined as trial was closed by sponsor prior to meeting this objective
Time Frame: not analyzed
Population: Data could not be reported in the data table as the data were not collected due to study early termination.
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 0

9. Secondary Outcome: Incidence and Severity of Acute and Chronic GVHD
Description: Incidence and severity of acute and chronic GVHD unable to be determined as trial was closed by sponsor prior to meeting this objective
Time Frame: not analyzed
Population: Data could not be reported in the data table as the data were not collected due to study early termination.
Arm/Group | Pevonedistat and Azacitidine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: completion of Cycle 5 day 9, up to 1 year.
Arm/Group | Pevonedistat and Azacitidine
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pevonedistat and Azacitidine (N=2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pevonedistat and Azacitidine (N=2)
abdominal pain (Gastrointestinal disorders) | 1 (1)
activated partial thromboplastin (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
anemia (Blood and lymphatic system disorders) | 2 (15)
anorexia (General disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Back pain (General disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorder (Blood and lymphatic system disorders) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Bruising (General disorders) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Investigations) | 2 (2)
Cytomegalovirus infection reactivation (Infections and infestations) | 2 (2)
Dizziness (General disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphasia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Edema trunk (General disorders) | 1 (1)
Ejection fraction decreased (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
Fecal incontinence (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Flank pain (Renal and urinary disorders) | 1 (1)
Gait disturbance (Nervous system disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperglycemia (Investigations) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Investigations) | 2 (4)
Hypermagnesemia (Investigations) | 1 (1)
Hypernatremia (Investigations) | 2 (2)
Hyperphosphatemia (Investigations) | 2 (2)
Hypertension (Cardiac disorders) | 2 (2)
Hyperuricemia (Investigations) | 2 (3)
Hypoalbuminemia (Investigations) | 2 (2)
Hypocalcemia (Investigations) | 2 (2)
Hyponatremia (Investigations) | 2 (4)
Hypophosphatemia (Investigations) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
INR increased (Blood and lymphatic system disorders) | 2 (2)
Lipase increased (Investigations) | 1 (1)
Localized edema (Cardiac disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (16)
Nail discoloration (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neck edema (General disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (19)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (General disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Sepsis (Infections and infestations) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1)
Sinus tachycardia (Blood and lymphatic system disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
White blood cell decreased (Blood and lymphatic system disorders) | 2 (18)

LIMITATIONS AND CAVEATS:
limitations to the data exist as the sponsor closed the study prior to subjects meeting study endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT03709576/Prot_SAP_000.pdf